CLINICAL TRIAL: NCT00556426
Title: The Bard® Recovery® Filter Registry (EVEREST) for Patients Who Are Candidates for an Optional (Retrievable) Inferior Vena Cava Filter That Undergo Placement of the Bard® Recovery® Filter.
Brief Title: Prospective, Multi-center, Single-arm Study to Assess the Safety of Retrieval of the Recovery G2 Filter.
Acronym: EVEREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-RC-1332
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Results first posted 2011-05-11 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Pulmonary Embolism; Venous Thromboembolic Disease
Keywords: Venous Thromboembolic Disease; IVC Filter; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Filter (Experimental): All subjects enrolled to the study are in this arm. All subjects receive a filter.
  Interventions: Device: Bard Recovery G2 Filter System

INTERVENTIONS:
Device: Bard Recovery G2 Filter System — Retrieval of previously placed RECOVERY G2 IVC filter
  Other Names: Bard Recovery G2 Filter

SUMMARY:
This study was designed to assess the safety of retrieval of the Bard Recovery® G2® Filter System. The G2 filter is an FDA-cleared device for inferior vena caval interruption in patients with pulmonary thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at temporary , increased risk of pulmonary embolism requiring caval interruption

Exclusion Criteria:

* The patient has implanted filter in the IVC or superior vena cava (SVC)
* The patient has a duplicated or left-sided IVC
* The patient has a known untreatable or uncontrollable malignancy
* The patient has severe spinal deformity
* The patient has a creatinine > 2.0 mg/dl
* The patient has a life expectancy of < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Kaufman, MD, Principal Investigator — OHSU, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven Investigators at 11 sites enrolled a total of 100 study subjects between December 7, 2005 and July 24, 2006.
Groups:
- All Patients Receiving the Filter: All enrolled subjects
Period: Overall Study
Arm/Group | All Patients Receiving the Filter
Started | 100
Completed | 91
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving a Filter: Patients who were at temporary, increased risk of pulmonary embolism requiring inferior vena cava (IVC) interruption, and for whom Recovery G2 Filter retrieval could reasonably be expected to occur within 6 months of device placement.
Arm/Group | Participants Receiving a Filter
Number analyzed (Participants) | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 67
Region of Enrollment [Number; unit: participants]
  United States | 100
Indication for Placement [Number; unit: Number of Participants] — Patients with active thromboembolic disease (the presence of Deep Vein Thrombosis (DVT) or pulmonary embolism (PE) within 3 months of study enrollment).
  Number of Participants
    active thromboembolic disease | 43
    no active thromboembolic disease | 57

OUTCOME MEASURES:

1. Primary Outcome: Technical Success (Retrieval)
Description: Technical success for retrieval of the filter such that the entire filter is removed.
Time Frame: 1 month post filter retrieval or through 6 months following implantation
Population: 61 of 100 patients enrolled underwent filter retrieval during the study.
Measure: Number; unit: participants
Arm/Group | All Patients Receiving the Filter
Number analyzed (Participants) | 61
participants | 58

2. Primary Outcome: Clinical Success (Retrieval)
Description: technical success without subsequent damage to the cava wall or other retrieval-related complications requiring intervention.
Time Frame: Time of Retrieval or through 6 months of implantation
Population: 61/100 patients experienced filter retrieval during the study
Measure: Number; unit: participants
Arm/Group | All Patients Receiving the Filter
Number analyzed (Participants) | 61
participants | 57

3. Primary Outcome: Percentage of Participants With Adverse Events Through 30 Days Post Retrieval
Description: Adverse events occurring at the time of retrieval through 30 days post filter retrieval procedure
Time Frame: 30 days post retrieval
Population: 61 of 100 patients underwent filter retrieval during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients Receiving the Filter
Number analyzed (Participants) | 61
percentage of participants | 14.8 [7.1 to 26.6]

4. Secondary Outcome: Filter Migration > 2cm
Description: Percentage of subjects experiencing filter migrations from the initial placement position of 2cm or more.
Time Frame: 30 days post retrieval or 6 months following filter placement
Population: Migration measurement made for 58 retrieved subjects, 22 non-retrieved subjects reaching the 6 month visit, and 2 non-retrieved subjects with attempted retrievals and imaging.
Measure: Number; unit: Percent Subjects with Filter Migration
Arm/Group | All Patients Receiving the Filter
Number analyzed (Participants) | 82
Percent Subjects with Filter Migration | 12.2

5. Secondary Outcome: Incidence of Filter Fracture
Description: occurrence of fracture assessed at retrieval by the Investigator (broken filter arms, legs, or other components)
Time Frame: at 6 months or at retrieval of the filter
Population: adequate imaging was available to assess filter integrity in 83 of the 100 participants.
Measure: Number; unit: number of fractured filters
Groups:
- Fractured Filters: retrieval of the filter such that the entire filter is retrieved
Arm/Group | Fractured Filters
Number analyzed (Participants) | 83
number of fractured filters | 1

ADVERSE EVENTS:
Arm/Group | All Patients Receiving the Filter
Serious Adverse Events (participants affected / at risk) | 6/100
Other Adverse Events (participants affected / at risk) | 70/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Receiving the Filter (N=100)
Caval Stenosis (Vascular disorders) | 1 (76)
Deep Vein Thrombosis (Vascular disorders) | 1 (76)
Discomfort due to device penetration (General disorders) | 1 (76)
Inferior Vena Caval Occlusion (Vascular disorders) | 1 (76)
Pulomonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (76)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Receiving the Filter (N=100)
Abdominal Mass (Gastrointestinal disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Acute Psychosis (Psychiatric disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Adrenal Hemorrhage (Vascular disorders) | 1 (1)
Adverse Drug Reaction (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 15 (15)
Anemia Postoperative (Injury, poisoning and procedural complications) | 1 (1)
Anticoagulation Drug Level Above Therapeutic (Investigations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arterial Hemorrhage (Vascular disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Atrial Flutter (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Breast Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 3 (3)
Catheter Site Hemorrhage (Vascular disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Clostridium Colitis (Infections and infestations) | 3 (3)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Confusional State (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 13 (13)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Device Migration (Injury, poisoning and procedural complications) | 10 (10)
Diabetic Gastroparesis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dislocation of Joint Prosthesis (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Edema Peripheral (General disorders) | 2 (2)
Endocarditis Staphylococcal (Infections and infestations) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1)
Frequent Bowel Movements (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 3 (3)
Gastrointestinal Stenosis (Gastrointestinal disorders) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1)
Groin Abscess (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Heparin Induced Thrombocytopenia (General disorders) | 2 (2)
Hiatus Hernia (Gastrointestinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1)
Incision Site Complication (Injury, poisoning and procedural complications) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Joint Dislocation (Musculoskeletal and connective tissue disorders) | 2 (2)
Large Intestinal Ulcer Hemorrhage (Gastrointestinal disorders) | 1 (1)
Liver Function Test Abnormal (Investigations) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1)
Major Depression (Psychiatric disorders) | 4 (4)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1)
Micturition Urgency (Renal and urinary disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Obsessive Compulsive Disorder (Psychiatric disorders) | 1 (1)
Oral Candidiasis (Infections and infestations) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pain (General disorders) | 4 (4)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic Abscess (Infections and infestations) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Pericardial Hemorrhage (Cardiac disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Infections and infestations) | 12 (12)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postmastectomy Lymphedema (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Infection (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Pyuria (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Renal Cysts (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 3 (3)
Renal Impairment (Renal and urinary disorders) | 2 (2)
Renal Mass (Renal and urinary disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Restless Leg Syndrome (Nervous system disorders) | 1 (1)
Retroperitoneal Hematoma (Gastrointestinal disorders) | 1 (1)
Scan Adrenal Gland Abnormal (Investigations) | 1 (1)
Scrotal Edema (Reproductive system and breast disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 4 (4)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 12 (12)
Vena Cava Thrombosis (Vascular disorders) | 1 (1)
Vena Caval Injury (Vascular disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 3 (3)
Viral Infection (Infections and infestations) | 1 (1)
Vocal Cord Paresis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days